CLINICAL TRIAL: NCT03526523
Title: Testing the Efficacy of Mindfulness-based Stress Reduction as a Prophylactic Intervention in the Prevention of Perimenopausal Depression: a Randomized Trial
Brief Title: Testing the Efficacy of Mindfulness-based Stress Reduction in the Prevention of Perimenopausal Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Regina (Other)
Collaborators: Saskatchewan Health Research Foundation (Other); Saskatchewan Centre for Patient-Oriented Research (Other); University of Calgary (Other); Saskatchewan Health Authority - Regina Area (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: REB #2018-050
Record Dates: First submitted 2018-05-03; First posted 2018-05-16 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2020-12

CONDITIONS: Perimenopausal Depression; Depressive Symptoms
Keywords: Mindfulness based stress reduction; Perimenopausal depression; Menopause transition
MeSH Terms: conditions — Depression | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Intervention Model Description: A stratified randomization method will be used to balance the number of baseline stressful life events in each treatment group (<3 vs. 3+ in the last 6 months). Randomization will be performed once baseline stressful life events are determined.
Who Masked: Outcomes Assessor
Masking Description: The staff member who will be assessing for the presence of major depressive disorder in the follow-up period (in cases where a participant's CES-D score is 16 or greater) will be unaware of the participant's treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Treatment (Experimental): Mindfulness-based stress reduction
  Interventions: Behavioral: Mindfulness-based stress reduction
- Waitlist control (No Intervention): The active treatment will be received only after the outcomes monitoring period is complete.

INTERVENTIONS:
Behavioral: Mindfulness-based stress reduction — 8 weekly 2.5-hour group sessions of mindfulness based stress reduction, led by a certified MBSR instructor
  Arms: Active Treatment

SUMMARY:
Depression is the leading cause of disability worldwide and a risk factor for other diseases. While women are at elevated risk for depression in general, the menopause transition is a particularly vulnerable time for many women, with the risk for depression increasing 2-4 fold. The objective of this research study is to determine whether mindfulness-based stress reduction (MBSR), an 8-week structured intervention involving meditation and yoga, has any beneficial mood effects for women undergoing this vulnerable time.

DETAILED DESCRIPTION:
The menopause transition (a.k.a. perimenopause) represents the reproductive stage transitioning from regular menstrual cycles through the loss of ovulatory function and to the complete cessation of menses. The latter marks the onset of menopause. All middle-aged women experience the menopause transition, which, on average, extends 5-6 years surrounding the last menstrual period. In Saskatchewan, roughly 80 000 women are currently of perimenopausal age. An estimated 26-33% of women develop clinically significant depressive symptoms during the perimenopause. Rates of diagnosed major depressive disorder during the menopause transition range between 12 and 23%. Mounting evidence findings from the PI and others suggests that the erratic fluctuations in estradiol that occur during the normal menopause transition play a key role. Specifically, increased estradiol fluctuation may increase one's sensitivity to stress both in the laboratory and in the context of real-world stressful life events, resulting in an increased risk for clinically significant depressive symptoms.

MBSR has proven to be very effective at increasing stress resilience and improving emotional wellbeing in a variety of populations. Thus, in the current SHRF-funded project, we will examine the prophylactic mood benefits of MBSR. We hypothesize that MBSR will increase women's resilience in the context of stress-sensitizing hormonal fluctuation in the menopause transition, making them less prone to developing depressive symptoms.

The current project will be composed of five components: 1) Enrollment session; 2) Hormonal Sensitivity Assessment (1 month); 3) Treatment Phase (8 weeks); 4) Follow-Up Phase (6 months) and 5) Waitlist Control Group Treatment (8 weeks). Each component is described in detail below:

1. Enrollment Session. After completing an eligibility screening over the phone, a trained research assistant (RA) will conduct an enrollment session over the phone with the prospective participant. The participant will be emailed a Powerpoint presentation summarizing the study and a link to a Qualtrics survey that will contain an electronic version of the consent form. Over the phone, the RA will review the Powerpoint slides and consent form. Once consent is obtained, the RA will administer the Structured Clinical Interview for the Diagnostic and Statistical Manual of Mental Disorders-5 (SCID-RV) for axis I disorders to screen for the presence of current psychiatric disorders as well as assess past major depressive episodes. The participant will then follow the RA's instructions on how to download the Expimetrics application on their smart phone, which they will use to complete study component #2 (described below). After the phone call, participants will be emailed a link to a Qualtrics survey containing a number of questionnaires assessing demographic information as well as psychological variables that may predict participant outcomes. The RA will instruct the participant to complete the survey at their convenience over the following 7 days. The RA will also mail a kit containing 12 2-ml vials contained in a small cardboard box and 10 ovulation predictor tests. Next, participants will complete an electronic version of a number of questionnaires, described below, with the use of Qualtrics. Finally, participants will be given instructions on how to take an ovulation test and how to collect urine samples at home.
2. Hormonal Sensitivity Assessment (1.5 months). Starting on the first day of their next menstrual period following the enrolment session, participants will complete the Daily Rating of Severity of Problems (DRSP) for approximately 45 days (if possible, using the Expimetrics smart phone app). Starting on day seven of their menstrual cycle, they will take an ovulation predictor test upon waking each day until a positive test is obtained (usually 6-8 days). Once a positive test is obtained, the participant will notify a research assistant by text, email or phone. In addition, they will be asked to collect a small sample of urine every other day for 30 days. The DRSP should be completed daily until the last day of urine collection.
3. MBSR Intervention (8 weeks). The intervention is provided over the course of eight weekly 150-minute sessions and one 7-hour weekend intensive silent retreat. The MBSR program, modeled after the work of Jon Kabat-Zinn and colleagues at the Stress Reduction and Relaxation Clinic-Massachusetts Medical Center, has been used and adapted by Dr. Campbell and his colleagues at the University of Calgary for numerous populations. The MBSR program consists of three primary components: 1) theoretical material related to relaxation, meditation, and the body-mind connection, 2) experiential practice of meditation and yoga during the group meetings and home based practice, and 3) group process focused on problem solving related to impediments to effective practice, practical day-to-day applications of mindfulness, and supportive interaction between group members. A booklet is distributed containing information pertinent to each week's instruction, including a bibliography for those wishing to pursue relevant themes in greater depth, and 2 CDs with guided meditation to help with home practice. Each week, participants will be asked to record all between-session home practice.

   All sessions will be audiotaped; audiotapes will be randomly selected to be viewed by Dr. Campbell to monitor treatment fidelity. After evaluating the tapes, both written and verbal feedback will be provided to the instructor to support compliance with the treatment protocol. Note that audiotapes will not reveal the identity of any of the participants.
4. Follow-up Period (6 months). Immediately following the intervention and every two weeks for 6 months, participants from both treatment groups will be emailed a link to a Qualtrics survey including the CES-D. The following questionnaires will also be included in the survey immediately following the intervention as well as months 2, 4 and 6: the Perceived Stress Scale, the State-Trait Anxiety Inventory, the Five Facet Mindfulness Questionnaire and the Connor-Davidson Resilience Scale. For participants without an email address, an RA will complete the survey with them over the phone. Participants obtaining a CES-D score ≥16 will be contacted by an RA to complete the mood module of the SCID-5 over the phone to identify cases of major depression. Importantly, all post-randomization correspondence with participants will be carried out by staff members who are blinded to participants' treatment condition.
5. Waitlist MBSR Intervention (8 weeks). Following the six-month follow-up, members of each wave's waitlist control group will receive the MBSR intervention. Although this will serve no research purpose, we believe offering MBSR to all participants, rather than using a "no treatment" condition will make the trial more equitable and appealing.

ELIGIBILITY:
Inclusion Criteria:

* in the early or late menopause transition according to the Stages of Reproductive Aging Workshop (STRAW+10) criteria, defined as menstrual cycle length 7+ days shorter or longer than usual or the presence of amenorrhea lasting 60 days or more (but less than 12 months)

Exclusion Criteria:

* current psychiatric diagnosis of major depressive disorder, bipolar disorder, a psychotic disorder or any other psychiatric diagnosis rated "severe" based on DSM-5 criteria
* use of medications affecting mood (e.g. antidepressants) or ovarian hormone levels (e.g. oral contraceptives)
* pregnant or nursing
* currently receiving a psychological treatment for depression
* major life-threatening health conditions.

Ages: 42 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 104 (Actual)
Dates: Start 2018-07-05 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-03-20 (Actual)

PRIMARY OUTCOMES:
Depressive symptoms | 6 months (CES-D completed every 2 weeks)
  Mean score on the Center for Epidemiologic Studies Depression Scale (CES-D), which assesses depressive symptoms. Total scores can range from 0 to 60, with a higher score indicating more severe symptoms.

SECONDARY OUTCOMES:
Occurrence of elevated depressive symptoms (ordinal) | 6 months (CES-D completed every 2 weeks)
  Number of times a participant obtains a score of 16 or above on the Center for Epidemiologic Studies Depression Scale (CES-D), which assesses depressive symptoms. Total scores can range from 0 to 60, with a higher score indicating more severe symptoms.
Occurrence of elevated depressive symptoms (binary) | 6 months (CES-D completed every 2 weeks)
  Whether or not a participant obtains a score of 16 or above on the Center for Epidemiologic Studies Depression Scale (CES-D) at least once. The CES-D assesses depressive symptoms. Total scores can range from 0 to 60, with a higher score indicating more severe symptoms.
Occurrence of major depressive episodes | 6 months (SCID is administered in instances where a score of 16 or above is obtained on the Center for Epidemiologic Studies Depression Scale)
  Whether or not a participant meets all 5 criteria for a major depressive episode according to the Structured Clinical Interview for the Diagnostic and Statistical Manual of Mental Disorders-5 (SCID-5).

OTHER OUTCOMES:
Perceived stress | 6 months (PSS is completed at months 0, 2, 4 and 6)
  Mean score on the Perceived Stress Scale (PSS). Scores range from 0 to 40, with higher scores indicating greater perceived stress.
Stress resilience | 6 months (completed at months 0, 2, 4 and 6)
  Mean score on the Connor-Davidson Resilience Scale, which assesses resilience to stress. Scores range from 0 to 100, with higher scores indicating greater resilience.
Trait Anxiety | 6 months (completed at months 0, 2, 4 and 6)
  Mean score on Form Y of the State-Trait Anxiety Inventory, which assesses trait anxiety. Scores range from 20 to 80, with higher scores indicating greater anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Gordon, PhD, Principal Investigator — University of Regina
Locations (1):
- University of Regina, Department of Psychology, Regina, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oldenhave A, Jaszmann LJ, Haspels AA, Everaerd WT. Impact of climacteric on well-being. A survey based on 5213 women 39 to 60 years old. Am J Obstet Gynecol. 1993 Mar;168(3 Pt 1):772-80. doi: 10.1016/s0002-9378(12)90817-0. PMID 8456878
- [Background] Treloar AE. Menstrual cyclicity and the pre-menopause. Maturitas. 1981 Dec;3(3-4):249-64. doi: 10.1016/0378-5122(81)90032-3. PMID 7334935
- [Background] Avis NE, McKinlay SM. The Massachusetts Women's Health Study: an epidemiologic investigation of the menopause. J Am Med Womens Assoc (1972). 1995 Mar-Apr;50(2):45-9, 63. PMID 7722206
- [Background] Bromberger JT, Kravitz HM, Chang YF, Cyranowski JM, Brown C, Matthews KA. Major depression during and after the menopausal transition: Study of Women's Health Across the Nation (SWAN). Psychol Med. 2011 Sep;41(9):1879-88. doi: 10.1017/S003329171100016X. Epub 2011 Feb 9. PMID 21306662
- [Background] Bromberger JT, Matthews KA, Schott LL, Brockwell S, Avis NE, Kravitz HM, Everson-Rose SA, Gold EB, Sowers M, Randolph JF Jr. Depressive symptoms during the menopausal transition: the Study of Women's Health Across the Nation (SWAN). J Affect Disord. 2007 Nov;103(1-3):267-72. doi: 10.1016/j.jad.2007.01.034. Epub 2007 Feb 28. PMID 17331589
- [Background] Cohen LS, Soares CN, Vitonis AF, Otto MW, Harlow BL. Risk for new onset of depression during the menopausal transition: the Harvard study of moods and cycles. Arch Gen Psychiatry. 2006 Apr;63(4):385-90. doi: 10.1001/archpsyc.63.4.385. PMID 16585467
- [Background] Freeman EW, Sammel MD, Liu L, Gracia CR, Nelson DB, Hollander L. Hormones and menopausal status as predictors of depression in women in transition to menopause. Arch Gen Psychiatry. 2004 Jan;61(1):62-70. doi: 10.1001/archpsyc.61.1.62. PMID 14706945
- [Background] Woods NF, Smith-DiJulio K, Percival DB, Tao EY, Mariella A, Mitchell S. Depressed mood during the menopausal transition and early postmenopause: observations from the Seattle Midlife Women's Health Study. Menopause. 2008 Mar-Apr;15(2):223-232. doi: 10.1097/gme.0b013e3181450fc2. PMID 18176355
- [Background] Bromberger JT, Kravitz HM, Wei HL, Brown C, Youk AO, Cordal A, Powell LH, Matthews KA. History of depression and women's current health and functioning during midlife. Gen Hosp Psychiatry. 2005 May-Jun;27(3):200-8. doi: 10.1016/j.genhosppsych.2005.01.007. PMID 15882767
- [Background] Pratt LA, Brody DJ. Depression in the United States household population, 2005-2006. NCHS Data Brief. 2008 Sep;(7):1-8. PMID 19389321
- [Background] Gordon JL, Eisenlohr-Moul TA, Rubinow DR, Schrubbe L, Girdler SS. Naturally Occurring Changes in Estradiol Concentrations in the Menopause Transition Predict Morning Cortisol and Negative Mood in Perimenopausal Depression. Clin Psychol Sci. 2016 Sep;4(5):919-935. doi: 10.1177/2167702616647924. PMID 27867758
- [Background] Gordon JL, Rubinow DR, Eisenlohr-Moul TA, Leserman J, Girdler SS. Estradiol variability, stressful life events, and the emergence of depressive symptomatology during the menopausal transition. Menopause. 2016 Mar;23(3):257-66. doi: 10.1097/GME.0000000000000528. PMID 26529616
- [Background] Freeman EW, Sammel MD, Lin H, Nelson DB. Associations of hormones and menopausal status with depressed mood in women with no history of depression. Arch Gen Psychiatry. 2006 Apr;63(4):375-82. doi: 10.1001/archpsyc.63.4.375. PMID 16585466